CLINICAL TRIAL: NCT00378300
Title: Probiotics Ameliorate Atopic Dermatitis by Induction of T Regulatory Cells
Brief Title: The Effects of Probiotics in Atopic Dermatitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funding to support this fellow-in-training initiated study.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Michael Land, UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-08-007-01
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Probiotics; T Regulatory Cells
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Oral Probiotics

SUMMARY:
The purpose of this study is to study the clinical effects of taking probiotics in patients who have moderate to severe atopic dermatitis. There has been several studies showing improvement in the severity of atopic dermatitis after taking probiotics. The mechanism of this improvement is currently unknown. We propose that probiotics improve atopic dermatitis by stimulating, or increasing, the activity of a special type of cell called the T Regulatory cell--which can suppress the activity of allergic disease.

DETAILED DESCRIPTION:
The central hypothesis of this study is that a subset of commercially available probiotic formulations will ameliorate moderate to severe atopic dermatitis in children by inducing the development of T Regulatory (Treg) cells. We specifically hypothesize that the probiotic mixture that induces Treg activity in vitro, will also improve the severity of atopic dermatitis in a specific patient by inducing Treg activity in vivo.

1. We will determine whether probiotic mixtures are better able to ameliorate the severity of atopic dermatitis when compared to patients treated with placebo. We will conduct a 4-week randomized, double-blind, placebo controlled clinical trial designed to evaluate the efficacy of probiotics in reducing the clinical severity of atopic dermatitis as assessed by our primary outcome measure, the SCORing Atopic Dermatitis (SCORAD) index. We specifically hypothesize that probiotics will clinically improve the disease.
2. We will assess whether probiotic mixtures induce the development of T regulatory cells in patients with atopic dermatitis.

A. We will measure the relative levels of Tregs in peripheral blood before and after probiotic or placebo administration in order to assess whether the probiotic mixtures alter Treg development in vivo, and whether these changes correlate with improvement in clinical scores. Primary outcomes will be measurements of gene expression and absolute increases in cell population. We specifically hypothesize that probiotics will increase Treg activity.

B. We will also determine if all patients' Tregs have in vitro responses to probiotics. This data will be used to correlate whether clinical responders in the study also have strong in vitro responses.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months to 3 years
* Physician diagnosis of moderate to severe atopic dermatitis as defined by the Hanifin and Rajka criteria
* Ability to take enterally commercially available probiotics by powder form added to food or drink
* Ability to undergo venipuncture or dermal puncture (if less than 1 year old)

Exclusion Criteria:

* Prior exposure to probiotics
* Current antibiotic administration
* Known history of chronic medical condition such as congenital heart disease, liver or kidney disease, or immune deficiency
* Absence of T regulatory cell induction by probiotic bacteria on initial laboratory assessment
* Any other condition in which the Investigators involved in the study determine potential subject is unsuitable for the study

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
SCORAD Score change taken at baseline and after 1 month of either probiotic or placebo
T Regulatory cell activity change taken at baseline and after 1 month of either probiotic or placebo

SECONDARY OUTCOMES:
Dermatitis Family Impact Questionnaire change taken at baseline and after 1 month of either probiotic or placebo
T Regulatory cell activity when exposed to probiotics in vitro
Change in Serum IgE or IgG levels taken at baseline and after 1 month of either probiotic or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Land, MD, Principal Investigator — University of California, Los Angeles; Martin G Martin, MD, MPP, Principal Investigator — University of California, Los Angeles; Robert L Roberts, MD, PhD, Principal Investigator — University of California, Los Angeles; Tatiana Hernandez, Study Director — University of California, Los Angeles
Locations (1):
- UCLA Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Kalliomaki M, Salminen S, Arvilommi H, Kero P, Koskinen P, Isolauri E. Probiotics in primary prevention of atopic disease: a randomised placebo-controlled trial. Lancet. 2001 Apr 7;357(9262):1076-9. doi: 10.1016/S0140-6736(00)04259-8. PMID 11297958
- [Background] Isolauri E, Arvola T, Sutas Y, Moilanen E, Salminen S. Probiotics in the management of atopic eczema. Clin Exp Allergy. 2000 Nov;30(11):1604-10. doi: 10.1046/j.1365-2222.2000.00943.x. PMID 11069570
- [Background] Pessi T, Sutas Y, Hurme M, Isolauri E. Interleukin-10 generation in atopic children following oral Lactobacillus rhamnosus GG. Clin Exp Allergy. 2000 Dec;30(12):1804-8. doi: 10.1046/j.1365-2222.2000.00948.x. PMID 11122221
- [Background] Kalliomaki M, Salminen S, Poussa T, Arvilommi H, Isolauri E. Probiotics and prevention of atopic disease: 4-year follow-up of a randomised placebo-controlled trial. Lancet. 2003 May 31;361(9372):1869-71. doi: 10.1016/S0140-6736(03)13490-3. PMID 12788576
- [Background] Rosenfeldt V, Benfeldt E, Nielsen SD, Michaelsen KF, Jeppesen DL, Valerius NH, Paerregaard A. Effect of probiotic Lactobacillus strains in children with atopic dermatitis. J Allergy Clin Immunol. 2003 Feb;111(2):389-95. doi: 10.1067/mai.2003.389. PMID 12589361
- [Background] Weston S, Halbert A, Richmond P, Prescott SL. Effects of probiotics on atopic dermatitis: a randomised controlled trial. Arch Dis Child. 2005 Sep;90(9):892-7. doi: 10.1136/adc.2004.060673. Epub 2005 Apr 29. PMID 15863468
- [Background] Viljanen M, Savilahti E, Haahtela T, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Kuitunen M. Probiotics in the treatment of atopic eczema/dermatitis syndrome in infants: a double-blind placebo-controlled trial. Allergy. 2005 Apr;60(4):494-500. doi: 10.1111/j.1398-9995.2004.00514.x. PMID 15727582
- [Background] Smits HH, Engering A, van der Kleij D, de Jong EC, Schipper K, van Capel TM, Zaat BA, Yazdanbakhsh M, Wierenga EA, van Kooyk Y, Kapsenberg ML. Selective probiotic bacteria induce IL-10-producing regulatory T cells in vitro by modulating dendritic cell function through dendritic cell-specific intercellular adhesion molecule 3-grabbing nonintegrin. J Allergy Clin Immunol. 2005 Jun;115(6):1260-7. doi: 10.1016/j.jaci.2005.03.036. PMID 15940144